CLINICAL TRIAL: NCT05177770
Title: A Phase 2 Trial of SRF617 in Combination With AB928 (Etrumadenant) and AB122 (Zimberelimab) in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of SRF617 With AB928 (Etrumadenant) and AB122 (Zimberelimab) in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated for strategic reasons, not due to any safety concerns.
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry); Surface Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF617-201
Record Dates: First submitted 2021-12-05; First posted 2022-01-05 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Prostate Cancer
Keywords: mCRPC; metastatic castration-resistant prostate cancer; prostate cancer; CD-39; PD-1; A2a; A2b; SRF617; AB122; AB928; adenosine pathway; cancer; immunotherapy; phase 2; efficacy; checkpoint inhibitor; adenosine receptor antagonist
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRF617 in combination with etrumadenant and zimberelimab (Experimental): All patients will receive SRF617 administered in combination with etrumadenant (AB928) and zimberelimab (AB122).
  Interventions: Drug: SRF617; Drug: etrumadenant; Drug: zimberelimab

INTERVENTIONS:
Drug: SRF617 — SRF617 is a fully human antibody designed to inhibit the enzymatic activity of CD39.
Drug: etrumadenant — Etrumadenant is an A2aR and A2bR antagonist.
  Other Names: AB928
Drug: zimberelimab — Zimberelimab is a fully human anti-PD-1 monoclonal antibody.
  Other Names: AB122

SUMMARY:
This trial will look at the safety and preliminary efficacy of SRF617 in combination with etrumadenant and zimberelimab in patients with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a phase 2, open-label, safety and preliminary efficacy trial in patients with mCRPC using the combination of SRF617, etrumadenant (AB928), and zimberelimab (AB122).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Metastatic CRPC with castrate levels of testosterone (≤ 50 ng/dL or ≤ 1.7 nmol/L).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Progressed (by PSA or radiologic criteria) during or following treatment with a novel androgen receptor signaling inhibitor (ARSI, eg, abiraterone, enzalutamide, apalutamide, darolutamide), which may have been given for either hormone-sensitive prostate cancer or CRPC.
* Received 1 to 2 prior lines of taxane chemotherapy, unless the physician and patient believe the patient is medically ineligible or the patient refuses (ineligibility or refusal must be documented in the source documents).
* Progressed by PSA or radiologic criteria on or during last therapy for prostate cancer.
* Measurable or non-measurable disease as per radiographic evaluation. Lesions situated in a previously irradiated area are considered evaluable if progression has been demonstrated in such lesions since radiation.

  • Note: If disease is considered non-measurable, a minimum PSA of 1 ng/dL is required with at least 1 confirmed rise at a minimum of a 1-week interval.
* Adequate hematologic function, defined as absolute neutrophil count ≥ 1.5 × 109/L, hemoglobin ≥ 9.0 g/dL, and platelet count ≥ 100 × 109/L. Transfusions are permitted to meet hemoglobin and platelet criteria. However, the patient must have a stable hemoglobin level and platelet count for ≥ 2 weeks prior to dosing without transfusion.
* Adequate renal function, defined as serum creatinine clearance ≥ 30 mL/min per Cockcroft-Gault formula.
* Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (≤ 3 × ULN if elevated because of Gilbert's syndrome, and ≤ 2 × ULN for patients with known liver metastases).
* Aspartate aminotransferase and alanine aminotransferase < 2.5 × ULN (< 5 × ULN if liver metastases present).
* Prothrombin time (PT) or international normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless the patient is receiving anticoagulant therapy, in which case PT/INR or aPTT must be within therapeutic range of intended use of anticoagulants.

Exclusion Criteria:

* Currently participating in or has participated in a trial of an investigational device or has used an investigational device within 21 days before the first dose of study drug.
* Any component of small cell or neuroendocrine histology.
* Previously received an anti-CD39 antibody, anti-CD39 targeted therapy, or other agent targeting the adenosine pathway.
* Prior treatment with programmed death-ligand 1 (PD-L1)/programmed death receptor-1 (PD-1) inhibitors.
* Prior treatment with ≥ 3 lines of taxane chemotherapy administered as a single agent or as part of a combination regimen.
* Symptomatic or untreated brain metastases (including leptomeningeal metastases). Patients previously treated for brain metastases must be at least 4 weeks from completion of radiation treatment with follow-up imaging showing no progression.
* Current pneumonitis with or without steroid requirement or history of pneumonitis requiring steroids.
* Another malignancy other than prostate within 2 years of trial entry, except for those with a low risk of spreading or negligible risk of death such as non-melanoma skin cancer or Ta superficial bladder cancer.
* Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Medical conditions requiring chronic steroid (ie, > 10 mg/day of prednisone or its equivalent).

  • Note: Replacement therapy (eg, levothyroxine, insulin, or physiologic corticosteroid replacement therapy for thyroid, adrenal, or pituitary insufficiency) is allowed.
* Administration of a live attenuated vaccine within 6 weeks before the first dose of study drug.

  • Exception: Health Authority approved COVID-19 vaccines are permitted.
* Any gastrointestinal condition that would preclude the use of oral medications (eg, difficulty swallowing, nausea, vomiting, or malabsorption).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vienna Reichert, PhD, Study Chair — Coherus BioSciences
Locations (9):
- United States (7):
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Michigan Health System, Ann Arbor, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - UT Southwestern, Dallas, Texas
  - START South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - START Mountain Region, Utah Cancer Specialists, West Valley City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (2):
  - BC Cancer - The Vancouver Centre, Vancouver, British Columbia
  - Université de Montreal - Centre de Recherche du Centre Hospitalier de L'Université de Montreal (CRCHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 participants were enrolled. 1 participant discontinued due to an adverse event prior to the first dose and was therefore not included in the analyses. 15 participants received study treatment and were included in the analyses.
Groups:
- SRF617 + Etrumadenant + Zimberelimab: SRF617 was administered in combination with etrumadenant and zimberelimab in 28-day cycles according to the following dosing schedule:
  * SRF617 1400 milligrams (mg) intravenously (IV) every 2 weeks (q2) on Days 1 and 15
  * Etrumadenant 150 mg orally daily
  * Zimberelimab 480 mg IV every 4 weeks (q4) on Day 1
Period: Overall Study
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Started | 16
Received at Least 1 Dose of Study Drug (Safety Analysis Set) | 15
Completed (Completion was defined as completing the safety follow up visit.) | 10
Not Completed | 6
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event prior to dosing | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received any amount of study drug
Groups:
- SRF617 + Etrumadenant + Zimberelimab: SRF617 was administered in combination with etrumadenant and zimberelimab in 28-day cycles according to the following dosing schedule:
  * SRF617 1400 mg IV every q2 weeks on Days 1 and 15
  * Etrumadenant 150 mg orally daily
  * Zimberelimab 480 mg IV q4 weeks on Day 1
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Response was defined as Prostate-Specific Antigen (PSA) decline of ≥ 50% (PSA50) and/or radiographic objective response of Complete Response (CR) or Partial Response (PR) per Prostate Cancer Working Group 3 (PCWG3) Criteria. The number of participants with response shows participants with any one or combination of these response types.
  * CR: Disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to < 10 millimeters (mm) in short axis
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum of diameters
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: The Response-Evaluable Analysis Set is defined as all participants at Baseline who received study drug and had at least 1 post-Baseline response assessment or who discontinued the treatment phase because of radiographic or symptomatic disease progression (including death caused by disease progression) within 6 weeks (+ 2 week window) of the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 15
Participants | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious Adverse Events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From date of first dose until 90 days after the last dose of treatment (maximum treatment exposure: 168 days)
Population: The Safety Analysis Set included all participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 15
Participants | 15

3. Secondary Outcome: Number of Participants With Response Per PCWG3 Criteria
Description: The number of participants achieving CR or PR by PCWG3 criteria is reported:
  * CR: Disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to < 10 millimeters (mm) in short axis
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum of diameters
  * Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions from the smallest value on trial (including Baseline, if that is the smallest). The sum of diameters must also demonstrate an absolute increase of at least 5 mm. Or, the appearance of one or more lesions
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from first documented response (PSA50 and/or CR/PR) to documented disease progression as determined by applicable disease criteria, or documented death due to any cause, whichever occured first.
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with CR, PR, or SD lasting a minimum of 12 weeks by PCWG3 or PSA50 criteria.
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With PSA50 Response
Description: PSA50 response is defined as a confirmed PSA decrease from Baseline of 50% or more based on 2 consecutive assessments measured 3 to 4 weeks apart.
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- SRF617 + Etrumadenant + Zimberelimab: SRF617 was administered in combination with etrumadenant and zimberelimab in 28-day cycles according to the following dosing schedule:
  * SRF617 1400 mg IV every q2 weeks on Days 1 and 15
  * Etrumadenant 150 mg orally daily
  * Zimberelimab 480 mg IV q4 weeks on Day 1b.
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 15
Participants | 0

7. Secondary Outcome: Number of Participants With PSA Decline of ≥ 30% (PSA30) Response
Description: PSA30 response is defined as a confirmed PSA decrease from Baseline of 30% or more based on 2 consecutive assessments measured 3 to 4 weeks apart.
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to PSA Progression
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

9. Secondary Outcome: Radiographic Progression Free Survival (PFS)
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

10. Secondary Outcome: Landmark PFS Rate
Description: Landmark PFS was defined as the percentage of participants who have not developed PFS events of death or documented disease progression as determined by applicable disease criteria.
Time Frame: Months 6 and 12
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

11. Secondary Outcome: Maximum Observed Serum Concentration of SRF617 (Cmax)
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Groups:
- SRF617 + Etrumadenant + Zimberelimab: Participants received SRF617 administered in combination with etrumadenant and zimberelimab.
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

12. Secondary Outcome: Minimum Observed Serum Concentration of SRF617 Prior to Administration of Subsequent Dose (Cmin)
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs)
Time Frame: From the date of first dose administration to the end of treatment (maximum exposure: 168 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Symptomatic Skeletal Events (SSEs)
Description: Number of participants with SSEs per PCWG3 criteria, defined as symptomatic fracture, radiation or surgery to bone, or spinal cord compression, is reported.
Time Frame: From date of first dose until 90 days after the last dose of treatment (maximum treatment exposure: 168 days)
Population: The Safety Analysis Set included all participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
Number analyzed (Participants) | 15
Participants | 4

ADVERSE EVENTS:
Time Frame: From date of first dose until 90 days after the last dose of treatment (maximum treatment exposure: 168 days)
Description: The Safety Analysis Set included all participants who received any amount of study drug. Also included is 1 participant who discontinued due to an adverse event prior receiving study drug.
Arm/Group | SRF617 + Etrumadenant + Zimberelimab
All-Cause Mortality (participants affected / at risk) | 4/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRF617 + Etrumadenant + Zimberelimab (N=16)
Spinal cord compression (Nervous system disorders) | 2 — Resulted in death of 1 participant
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1 — Resulted in death
Disease progression (General disorders) | 1 — Resulted in death
Cytokine release syndrome (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1 — Resulted in death
Back pain (Musculoskeletal and connective tissue disorders) | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 — Screen failure; discontinued prior to receiving study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRF617 + Etrumadenant + Zimberelimab (N=16)
Fatigue (General disorders) | 6
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
General physical health deterioration (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Oral dysaesthesia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Oesophageal pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Weight decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Lipase increased (Investigations) | 2
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Anosmia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hypoglossal nerve disorder (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Soft tissue infection (Infections and infestations) | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Eyelid function disorder (Eye disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4

LIMITATIONS AND CAVEATS:
This study was originally intended to be conducted in 2 stages (1 and 2); however, a strategic decision was made to terminate the study during Stage 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT05177770/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT05177770/SAP_001.pdf